CLINICAL TRIAL: NCT00888602
Title: An Open Label, Randomized, 4-Period Cross-over Study to Evaluate the Effects of Psyllium Taken Before a Meal on Postprandial Blood Glucose in Healthy Males
Brief Title: Study to Evaluate the Effects of Psyllium on Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2009001
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Healthy Men
MeSH Terms: interventions — Psyllium; Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MM1 - Meal (Experimental): 3.4g psyllium served with a meal
  Interventions: Dietary Supplement: 3.4 g psyllium
- MM2 - Meal (Experimental): 6.8 g psyllium served with a meal
  Interventions: Dietary Supplement: 6.8 g psyllium
- MM2 (no Meal) (Experimental): 6.8 g psyllium consumed with no meal
  Interventions: Dietary Supplement: 6.8 g psyllium
- Meal Only (Sham Comparator): meal only
  Interventions: Other: Meal

INTERVENTIONS:
Dietary Supplement: 3.4 g psyllium — 3.4 g psyllium served with meal
  Arms: MM1 - Meal
Dietary Supplement: 6.8 g psyllium — 6.8 g psyllium served with a meal
  Arms: MM2 - Meal
Dietary Supplement: 6.8 g psyllium — 6.8 g psyllium
  Arms: MM2 (no Meal)
Other: Meal — meal
  Arms: Meal Only

SUMMARY:
This is an open label, single use, randomized, 4-period cross-over study. In each period, subjects will receive one of 4 test combinations. Blood will be drawn prior to study product consumption and following study product consumption for glucose measures.

ELIGIBILITY:
Inclusion Criteria:

* male
* 18 to 50 years of age
* general good health
* Body Mass Index (BMI) in the range of 18.5-29.9 kg/m2
* fasting plasma blood glucose <126mg/dL
* not actively treated for high blood glucose
* willing and able to have blood drawn at multiple times during each 4 visits

Exclusion Criteria:

* history of allergy or hypersensitivity to inhaled or ingested psyllium or meal ingredients
* Phenylketonuria (PKU)
* an eating disorder
* following special medical or weight-loss dietary restrictions
* taking dietary supplements or prescription medication for the purpose of weight loss/management

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
to evaluate the effect of 2 dosing levels of psyllium on glucose in blood when taken prior to a meal vs. a meal alone | 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hill Top Research, Miamiville, Ohio, United States